CLINICAL TRIAL: NCT04162262
Title: Immediate and 12-week Effects of Exercise Versus Exercise and Instrument-Assisted Soft Tissue Mobilization for Plantar Fasciopathy Treatment: A Randomized Controlled Trial
Brief Title: Effects of Exercise Versus Exercise and Instrument-Assisted Soft Tissue Mobilization for Plantar Fasciopathy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L19-147
Record Dates: First submitted 2019-11-01; First posted 2019-11-14 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Plantar Fascitis
Keywords: Plantar Fascitis; Instrument-assisted soft tissue mobilization; Stretch and strengthening exercise; Plantar fasciopathy

STUDY DESIGN:
Intervention Model Description: This study is divided into two parts. Part I is a parallel-group, pre-test post-test randomized controlled superiority trial comparing the effects of stretching and strengthening exercises (SS) (Group 1) versus SS plus IASTM (SS+IASTM, Group 2) in subjects with PF. Outcomes will be assessed by a blinded investigator after one visit and 4, 8, and 12 weeks of treatment. Part II is a pre-test, posttest comparison of the short-term effects of IASTM on PF (Group 2) and control (Group 3) groups.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Random group allocation into Groups 1 and 2 will be performed using a 1:1 allocation ratio with permuted block sizes of 2 to 6. The investigators responsible for the weekly progression of the stretching and strengthening exercise protocol and the outcome assessor will be masked to the participants' assigned groups. The investigators providing instrument-assisted soft tissue mobilization will not be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stretching, Strengthening, and IASTM (Experimental): This group will attend eight weekly sessions, which will include initial screening tests and exercise education on visit 1 and strengthening and stretching exercise progression on visits 1-8. Data measurements will occur at weeks 0, 4, 8, and 12. This group will perform a 5-minute, self-paced warmup on a stationary bicycle followed by a 10-minute IASTM treatment. Test measurements will be performed before and immediately following the warmup and IASTM treatment. They will then perform stretching and strengthening exercises under the supervision of an investigator masked to treatment group weekly for eight visits. Exercise resistance will be increased as needed each week. In addition, participants will perform daily stretching and strengthening exercises at home.
  Interventions: Other: Instrumental-assisted soft tissue mobilization (IASTM); Other: High-Load Strength Training; Other: Plantar Flexor and Gastrocnemius Stretching
- Strengthening and Stretching (Active Comparator): This group will attend eight weekly sessions, which will include initial screening tests and exercise education on visit 1 and strengthening and stretching exercise progression on visits 1-8. Data measurements will occur at weeks 0, 4, 8, and 12. To equalize visit time with the Stretching, Strengthening, and IASTM group, subjects will perform 15 minutes of self-paced bicycle riding at the beginning of each session. They will then perform stretching and strengthening exercises under the supervision of an investigator masked to treatment group weekly for eight visits. Exercise resistance will be increased as needed each week. In addition, participants will perform daily stretching and strengthening exercises at home.
  Interventions: Other: High-Load Strength Training; Other: Plantar Flexor and Gastrocnemius Stretching
- Pain-free Comparison Group (Other): The third group is a pain-free comparison group. This group will come to the laboratory once. They will perform a 5-minute, self-paced warmup on a stationary bicycle followed by a 10-minute IASTM treatment. Test measurements will be performed before and immediately following the warmup and IASTM treatment. These measurements will be compared to the same measures from the Stretching, Strengthening, and IASTM group to examine outcome measure differences in those with and without plantar fasciopathy following a single IASTM treatment.
  Interventions: Other: Instrumental-assisted soft tissue mobilization (IASTM)

INTERVENTIONS:
Other: Instrumental-assisted soft tissue mobilization (IASTM) — Instrumental-assisted soft tissue mobilization (IASTM) will consist of treatment focused on the plantar surfaces of foot, posterior heel, and lower leg. The IASTM will be implemented using Graston Technique Instruments by clinicians trained and certified in the technique. Each 10-minute treatment will consist of two phases: 1) six-minute static phase, which includes tissue status screening and soft tissue mobilization, and 2) four-minute dynamic tissue mobilization phase. The treatment will focus on the web spaces of each toe plantarly, the metatarsal heads, the spaces between metatarsals, the medial and lateral plantar fascia borders, plantar fascia proximal origin, the heel, and the lower leg muscle groups. The targeted soft tissues are the plantar fascia, ankle plantar flexors, heel fat pad, Achilles tendon, and the gastrocnemius-soleus complex.
  Arms: Pain-free Comparison Group; Stretching, Strengthening, and IASTM
Other: High-Load Strength Training — Participants will perform a heel raise exercise used by Rathleff et al (2015). The exercise will be performed twice daily. While standing with the forefoot on a step, the toes will rest on a partially folded towel, placing them in a maximally dorsiflexed position. The exercise will consist of a maximum ankle plantar flexion followed by maximal dorsiflexion. The concentric plantar flexion and eccentric lowering phases will be 3 seconds, with a 2 second isometric pause in between. The exercise will be performed unilaterally if tolerated by the subject. Otherwise, a bilateral calf raise will be performed until the subject is able to perform the unilateral version. The exercise will be performed every other day and progressed throughout the trial as described by Rathleff and colleagues.
  Arms: Strengthening and Stretching; Stretching, Strengthening, and IASTM
Other: Plantar Flexor and Gastrocnemius Stretching — For the plantar flexor stretch (DiGiovanni et al, 2006), subjects will sit and cross the affected leg over the contralateral leg. Placing the affected side fingers on the plantar toes, distal to the metatarsophalangeal joints, they will passively dorsiflex the toes until they feel stretching in the arch of the foot. Subjects will be instructed to hold this stretch for 10 seconds and repeat it 10 times. The gastrocnemius stretch will be performed in supine with a towel placed around the distal foot and the foot actively inverted. With the knee extended, the subject will flex the hip while passively dorsiflexing the foot using the towel. This stretch will be held for 30 seconds and repeated 3 times. Subjects will be asked to perform both stretches three times each day.
  Arms: Strengthening and Stretching; Stretching, Strengthening, and IASTM

SUMMARY:
This study compares the addition instrument-assisted soft tissue mobilization (IASTM) to a program of home strengthening and stretching exercises to see whether adding weekly IASTM treatments improves plantar fasciopathy pain and plantar fascia stiffness.

DETAILED DESCRIPTION:
Plantar fasciopathy (PF) is the most common cause of inferior heel pain, and approximately 40% of patients report symptoms two years following initial diagnosis. Exercise therapy, including gastrocnemius and plantar fascia stretching, and high-load strengthening have been shown to improve plantar fascia pain and function; however, not everyone improves with these interventions, and they require several weeks or months to be effective. The addition of instrument-assisted soft tissue mobilization (IASTM) techniques may improve these outcomes. Moreover, shear wave elastography (SWE) is an imaging technology that may provide helpful information regarding PF diagnosis and prognosis. Therefore, research is required to investigate changes in plantar fascia stiffness following exercise and IASTM interventions.

This study is divided into two Parts. Part I is a parallel-group, pre-test post-test randomized controlled superiority trial comparing the long-term effects of stretching and strengthening exercises (SS) (Group 1, n=35) versus SS plus IASTM (SS+IASTM, Group 2, n=35) in subjects with PF. The study is approved by the local Intuitional Review Board. The Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines for reporting of randomized interventional trials will be followed. Exercise interventions will be reported according to the Consensus on Exercise Reporting Template (CERT) guideline. Part II is a pre-test, post-test comparison of the short-term effects of IASTM on PF. Subjects from Group 2 of Part I (n=35) and a age and sex-matched healthy comparison group (Group 3, n=35) will participate in Part II.

Random group allocation into SS and SS+IASTM Groups will be performed by an independent statistician using the R Statistics package using a 1:1 allocation ratio with permuted block sizes of 2 to 6. Although it is not possible to blind study participants, the investigators performing the weekly interventions and measurements will be blinded to the subjects' group allocation.

After randomization subjects will receive a booklet that describes their condition and contains exercise instructions and an exercise training and medication usage diary. Group 1 will receive a sheet listing evidence for the beneficial effects of stretching and high-load strengthening. Group 2 will additionally receive information regarding the hypothesized benefits of IASTM. After group allocation and reading the appropriate booklet, subjects will complete the Credibility/Expectancy Questionnaire (CEQ), which contains six items requiring subjects to rate the credibility of the intervention and their expectations.

Both groups will perform an identical exercise program but will additionally receive once weekly IASTM treatments over an 8-week period. The weekly and total treatment time in Groups 1 and 2 will be the same, 15 minutes/week for 8 weeks. Group 3 (Comparison Group) will be recruited in clusters of five after every 5 subjects are recruited into Group 2 (SS+IASTM) and will be matched to that group's age and BMI.

Overall, subjects in Groups 1 and 2 will visit the lab 10 times. First, they will attend eight weekly sessions, which will include initial screening tests and exercise education on visit 1, treatments according to group allocation on visits 1-8, and follow-up testing on visits 5, 9, and 10. Both groups will additionally perform daily stretching and strengthening exercises at home. Between sessions 9 and 10 (i.e., weeks 9-11), these subjects will be contacted via telephone for follow-up testing and encourage continued home exercise program compliance. Group 3 will attend one session. This session will include screening tests before and after one IASTM treatment.

Data will be summarized in descriptive statistics such as mean (standard deviation), median (interquartile range), and frequencies (percentage) as appropriate depending on the variable levels of measurement. Associations among categorical variables will be assessed using Chi-square or Fisher's exact test. Associations among continuous or ordinal level variables will be assessed using appropriate parametric or non-parametric correlation tests. Differences among demographic groups on continuous baseline variables will be assessed using t-test and ANOVA or their non-parametric alternatives (Mann-Whitney or Kruskal Wallis tests) where appropriate.

The examined data in this study are clustered (nested) in nature. For example, the Foot Health Status, a dependent variable which is measured for both groups (the SS and SS + IASTM) through different subscales including pain subscale, function subscale, footwear subscale, and general foot health subscale (level 1), at different time points (level 2), within each individual participant (level 3). Therefore, linear mixed modeling is a suitable analytical technique to handle the data and answer research questions.

Since the levels of the examined factors in the study constitute all the levels of interest for statistical inference, a covariance pattern fixed effects model that accounts for the covariance and correlational patterns among repeated measures could be the most suitable for this study to be utilized (among other different Mixed Model approaches that would be tested and implemented).

ELIGIBILITY:
Inclusion Criteria for Plantar Fasciopathy Groups

* age 18-60 years
* self-reported history of plantar heel pain for a minimum of 2 months prior to enrollment
* pain on palpation of the medial calcaneal tubercle or the proximal plantar fascia
* pain is worst when first standing or walking after rest
* willing to attempt not to use additional treatments (e.g., shoe modifications, foot orthoses/braces, injections, or surgery) during the trial period (12 weeks)
* willing to attempt to discontinue taking all pain-relieving medications except Tylenol or ibuprofen for plantar heel pain during the trial period (12 weeks).

Inclusion Criteria for Healthy Comparison Group:

* age and BMI matched with Group 2 subjects
* no history or symptoms of plantar heel pain in the past 12 months

Exclusion Criteria for all three groups:

* history of direct trauma to the foot with plantar fasciopathy
* inflammatory arthritis in the feet/ankle (e.g., ankylosing spondylitis or rheumatoid arthritis)
* metabolic or endocrine disorders (e.g., Type I or II diabetes)
* neurological disorders (e.g., Charcot-Marie-Tooth disease)
* prior foot surgery on the foot with plantar fasciopathy
* pregnancy (by self-report)
* corticosteroid injection to treat plantar fasciopathy in the past 12 weeks
* body mass index > 35 kg/m2
* receiving or applied for worker compensation benefits
* no physical activity above 5 (moderate activity) on a 10-point Rating of Perceived Exertion scale in the past 24 hours prior to the initial screening visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
The Foot Health Status Questionnaire Pain Subscale Score | Week 8
  This self-report questionnaire assesses individuals' foot health and function. The pain subscale evaluates type of pain and its severity and duration.

SECONDARY OUTCOMES:
Ankle range of motion | Baseline and weeks 4, 8, and 12
  Ankle dorsiflexion range of motion will be measured while the subject performs a weight-bearing lunge while facing a wall. Subjects will keep their heels on the ground and may keep contact on the wall in front of them with two fingers to maintain balance. The knee will be aligned with the second toe with the first toe 10 cm away from the wall. To perform the test, subjects will bring their knee forward towards the wall, keeping it aligned with the second metatarsal. If the knee contacts the wall while maintaining the heel on the ground, the foot will be moved back 1 cm at a time until the heel raises off the ground during the test performance. The final distance between the wall and the first toe will be recorded, and the test will be repeated three times.
First metatarsophalangeal range of motions | Baseline and weeks 4, 8, and 12
  First metatarsophalangeal (MTJ) joint range of motion will be measured using a 2D electrogoniometer (Noraxon Ultium, Scottsdale, AZ). The electrogoniometer will be placed along the ventral surface of the first metatarsal phalangeal joint. Subjects will stand with the feet shoulder-width apart. An investigator will lift the first toe and record dorsiflexion range of motion. No mid-foot or heel motion will be allowed during measurement. The range of motion will be measured three times.
Patient Acceptable Symptom State | Baseline and weeks 4, 8, and 12. Phone visits at weeks 9, 10, 11.
  Self-reported time to achieve a satisfactory result.
Credibility/Expectancy Questionnaire | Baseline visit
  Participants self-rate the credibility of the intervention and their expectations for recovery after they are informed of their group allocation but prior to any intervention.
Visual Analog Scale Pain Score | Baseline and weeks 4, 8, and 12.
  Heel pain severity on a 10-cm scale when getting out of bed in the morning
Plantar Fascia Shear Wave Velocity | week 0, 4, 8 and 12
  Ultrasound Shear Wave Elastography (Aixplorer, Axe-En-Provence, France, Version 10) will be used to measure plantar fascia shear wave velocity (m/s) at the 0.5 cm distal to the proximal calcaneal insertion and at the level of the navicular in the midfoot.
The Foot Health Status Questionnaire Footwear Subscale Score | Baseline and weeks 4, 8, and 12
  Evaluates lifestyle issues related to footwear and the feet.
The Foot Health Status Questionnaire General Foot Health Subscale Score | Baseline and weeks 4, 8, and 12
  Evaluates participants' self-perception of their feet.
The Foot Health Status Questionnaire Foot Function Subscale Score | Baseline and weeks 4, 8, and 12
  Evaluates the feet in terms of impact on physical function
Physical Activity Level | Baseline and weeks 4, 8, and 12
  Measured using the International Physical Activity Questionnaire short form (IPAQ), which estimates weekly physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Troy Hooper, PhD, Principal Investigator — Faculty
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT04162262/ICF_000.pdf